CLINICAL TRIAL: NCT03349593
Title: Prevalence of Hypovolemia and Heart Failure in Non-cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Myrberg, Principal investigator, Umeå University
Other Study IDs: 2016/361-31 II
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Hypovolemia; Heart Failure; Diastolic Dysfunction; Systolic Dysfunction; Venous; Return (Anomaly)
Keywords: Heart failure, diastolic dysfunction, venous return; Left ventricular filling pressures
MeSH Terms: conditions — Hypovolemia; Heart Failure; Congenital Abnormalities | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Preoperative transthoracic echocardiography

SUMMARY:
Prevalence of biventricular function of the heart and preoperative level of venous return is not known in non-cardiac non-morbid obese population.

The aim of the study is to assess the preoperative function of the heart and status of hypovolemia on the day of surgery.

DETAILED DESCRIPTION:
Preoperative transthoracic echocardiography (TTE) is conducted in 100 individuals. Biventricular function (i.e. systolic and diastolic properties), left ventricular filling pressures and level of venous return are assessed by TTE.

Moreover high-sensitive troponine I and Nt-proBNP, ECG are collected. Multiple echocardiographic parameters will be studied for feasibility in terms of preoperative assessment of the heart.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≤ 35 kg/m2, electively scheduled for breast cancer surgery, endocrinologic surgery (thyroid, parathyroid) and general abdominal surgery.

Exclusion Criteria:

* Not signed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Electively scheduled individuals for breast cancer surgery, endocrinologic surgery (thyroid, parathyroid) and general abdominal surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Hypovolemia | One hour before surgery
  Screening of preoperative level of venous return
Heart failure | One hour before surgery
  Screening of incidence of preoperative systolic and diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Tomi P Myrberg, MD PhD, Principal Investigator — Umeå University, Norrbotten county concil
Locations (1):
- Sunderby hospital, Luleå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stenberg Y, Rhodin Y, Lindberg A, Aroch R, Hultin M, Wallden J, Myrberg T. Pre-operative point-of-care assessment of left ventricular diastolic dysfunction, an observational study. BMC Anesthesiol. 2022 Apr 5;22(1):96. doi: 10.1186/s12871-022-01642-4. PMID 35382761